CLINICAL TRIAL: NCT07130188
Title: The Significance of Triglyceride Index and TG/HDL-C Ratios as Predictors of Acute Coronary Syndromes in Young Population and the Complexity of Coronary Artery Disease
Brief Title: Predictors for ACS and Complexity of CAD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Saleh Mohamed Saleh, Principal Investigator, Assiut University
Other Study IDs: Predictors for ACS
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: TG Index; TG/HDL-C Ratio; Young Population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PCI — Coronary angiography then SYNTAX score calculation

SUMMARY:
To evaluate the significance of the Triglyceride index and TG/HDL-C ratio as predictors of acute coronary syndromes in the young population

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains a major cause of morbidity and mortality worldwide, with a rising incidence of acute coronary syndromes (ACS) in young individuals under the age of 40. Early identification of at-risk individuals in this population is essential for implementing preventive strategies and reducing adverse outcomes【1,2】. Traditional risk factors such as hypertension, diabetes, smoking, and dyslipidemia are well-established; however, their predictive value in the young population is often limited【2】.

Recent studies have highlighted the significance of novel lipid-derived markers, particularly the triglyceride-glucose (TyG) index and the triglyceride-to-high-density lipoprotein cholesterol (TG/HDL-C) ratio, as potential predictors of insulin resistance, subclinical atherosclerosis, and cardiovascular events【1,3】. The TyG index and TG/HDL-C ratio are simple, cost-effective markers derived from routine laboratory parameters and have shown promising associations with metabolic syndrome, endothelial dysfunction, and coronary artery disease (CAD) severity【3,4】.

Despite emerging evidence in older adults, limited data exist regarding the utility of these markers in predicting ACS among the young population, where conventional risk scores often underestimate risk【4,5】. Early detection through these markers could improve risk stratification and guide preventive strategies.

This study aims to evaluate the significance of the TyG index and TG/HDL-C ratio as predictors of ACS in young adults, providing insight into their potential role in primary prevention

ELIGIBILITY:
Inclusion Criteria:

-

Age 18-40 years. Confirmed diagnosis of ACS (STEMI, NSTEMI). Willingness to participate with informed consent.

Exclusion Criteria:

* Age > 40 years old People with Previous ACS Patients known to have familial hyperlipidemia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adult patients (18-45 years) admitted with acute coronary syndrome (STEMI, NSTEMI) who undergo coronary angiography during index hospitalization. Patients must have fasting lipid profile and fasting glucose measured within 24 hours of admission. Exclusions include familial hyperlipidemia, chronic inflammatory/autoimmune disease, severe renal or liver failure, active infection, recent use of non-statin lipid-altering drugs, or missing data for TyG/TG-HDL-C calculation. Follow-up will be conducted at 12 and 36 months to assess outcomes.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Predictive value of TyG index and TG/HDL-C ratio for acute coronary syndrome (ACS) in young adults | On second day of admission
  Occurrence of ACS (defined as STEMI, NSTEMI confirmed by clinical assessment, ECG changes, and cardiac biomarkers according to accepted guideline criteria) and the diagnostic/predictive performance of baseline Triglyceride-glucose (TyG) index and TG/HDL-C ratio for ACS.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Mohamed Abdallah, Professor, Study Director — Assuit university - faculty of medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim MK, Ahn CW, Kang S, Nam JS, Kim KR, Park JS. Relationship between the triglyceride glucose index and coronary artery calcification in Korean adults. Cardiovasc Diabetol. 2017 Aug 23;16(1):108. doi: 10.1186/s12933-017-0589-4. PMID 28830471
- [Background] Khalaji A, Behnoush AH, Pasebani Y, Rafati A, Mahmoodi T, Arzhangzadeh A, Shamshiri Khamene S, MohammadKhawajah I, Mehrani M, Vasheghani-Farahani A, Masoudkabir F, Najafi K, Askari MK, Harrison A, Nelson JR, Hosseini K, Hernandez AV. Triglyceride-glucose index as a predictor of cardiac adverse events in acute coronary syndrome patients undergoing percutaneous coronary intervention: role of diabetes. BMC Cardiovasc Disord. 2024 Sep 27;24(1):514. doi: 10.1186/s12872-024-04191-5. PMID 39333881
- [Background] Liu Y, Zhu B, Zhou W, Du Y, Qi D, Wang C, Cheng Q, Zhang Y, Wang S, Gao C. Triglyceride-glucose index as a marker of adverse cardiovascular prognosis in patients with coronary heart disease and hypertension. Cardiovasc Diabetol. 2023 Jun 9;22(1):133. doi: 10.1186/s12933-023-01866-9. PMID 37296406
- [Background] Ren X, Chen ZA, Zheng S, Han T, Li Y, Liu W, Hu Y. Association between Triglyceride to HDL-C Ratio (TG/HDL-C) and Insulin Resistance in Chinese Patients with Newly Diagnosed Type 2 Diabetes Mellitus. PLoS One. 2016 Apr 26;11(4):e0154345. doi: 10.1371/journal.pone.0154345. eCollection 2016. PMID 27115999
- [Background] da Silva A, Caldas APS, Hermsdorff HHM, Bersch-Ferreira AC, Torreglosa CR, Weber B, Bressan J. Triglyceride-glucose index is associated with symptomatic coronary artery disease in patients in secondary care. Cardiovasc Diabetol. 2019 Jul 11;18(1):89. doi: 10.1186/s12933-019-0893-2. PMID 31296225